CLINICAL TRIAL: NCT03281005
Title: Calibration of Visual Function Evaluation Tests in Patients With Severe Vision Loss
Brief Title: Development of Visual Function Evaluation Method
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CRE170041
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2020-03

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis pigmentosa; Visual function evaluation
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Retinitis pigmentosa in Part 1A: Retinitis pigmentosa patients with severe visual impairment
- Retinitis pigmentosa in Part 1B: Retinitis pigmentosa patients with severe visual impairment
- Retinitis pigmentosa in Part 2: Retinitis pigmentosa patients with severe visual impairment
- Healthy volunteers in Part 3: Healthy volunteers

SUMMARY:
The objective of this study is to develop the comprehensive visual function evaluation method in severe visually impaired patient

DETAILED DESCRIPTION:
This study is a prospective observational study which consists of 4 Parts; Part 1A, 1B, 2 and 3. Part 1A has been conducted on 6 subjects diagnosed with retinitis pigmentosa. Additional examination will be performed using alternative devices imported outside Japan on subjects who completed Part 1A and re-consented (Part 1B). Based on the interim result of Part 1A, Part 2 will be conducted on another 6 subjects with retinitis pigmentosa with improved methodology and the devices used in Part 1B. Part 3 will be conducted in 6 healthy volunteers to obtain comparative data using devices used in Part 1B.

ELIGIBILITY:
Inclusion Criteria for patients with retinitis pigmentosa:

* Age: ≥ 20 years
* Subjects with severe visual disturbance (count-fingers or worse vision for severe eyes) at the time of obtaining the consent

Inclusion Criteria for healthy Volunteers:

* Age: ≥ 35 and ≤ 75 years
* Subjects with corrected visual acuity ≥ 1.0 with both eyes and without severe refractive error nor abnormal findings in slit-lamp microscopy, OCT, fundoscopy and pupillary function test at screening

Exclusion Criteria:

* Subjects who have participated in any other clinical trial or clinical study involving visual function evaluation within 6 months
* Subjects who have history of surgery, past history, and complications (cardiac/ hepatic/ renal/ respiratory/ hematological diseases, optic nerve diseases causing marked loss of visual field, and uveitis etc.) that potentially affect evaluation and safety of the study
* Pregnant women
* Subjects who are judged that continuation of the study is difficult during the study period
* Subjects who are employed by the company sponsoring this study, an organization or institution related to this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retinitis pigmentosa, healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Slit-lamp microscopy in Part 1A and 2 | Up to week 8
  To assess the visual function
Slit-lamp microscopy in Part 1B and 3 | Day 1
  To assess the visual function
Optical Coherence Tomography (OCT) test in Part 1A and 2 | Day 1
  To assess the visual function
Visual acuity test with Early Treatment Diabetic Retinopathy Study (ETDRS) in Part 1A and 2 | Up to week 8
  To assess the visual function
Visual acuity test with ETDRS in Part 1B | Day 1
  To assess the visual function
The 25-item National Eye Institute Visual Function Questionnaire (NEI VFQ-25) in Part 1A and 2 | Up to week 8
  To assess the visual function and the quality of life (QOL)
The 11-item National Eye Institute Visual Function Questionnaire (NEI VFQ-11) in Part 1A and 2 | Up to week 8
  To assess the visual function and QOL
Nottingham Adjustment Scale Japanese Version (NAS-J) in Part 1A and 2 | Up to week 8
  To assess the psychological adjustment
Daily living task dependent on vision (DLTV) in Part 1A and 2 | Up to week 8
  To assess QOL
Table test in Part 1A and 2 | Up to week 8
  To assess the visual function
Metropsis test in Part 1A and 2 | Up to week 8
  To assess the visual function
Low vision evaluator (LoVE) in Part 1A | Up to week 8
  To assess the visual function
White flash visual evoked potential (VEP) test in Part 1A and 2 | Up to week 8
  To assess the visual function
White flash VEP test in Part 1B and 3 | Day 1
  To assess the visual function
Color flash VEP test in Part 1A and 2 | Up to week 8
  To assess the visual function
Color flash VEP test in Part 1B and 3 | Day 1
  To assess the visual function
Electrically evoked response (EER) test in Part 1A and 2 | Up to week 8
  To assess the visual function
EER test in Part 1B and 3 | Day 1
  To assess the visual function
White flash electroretinography test in Part 1A, 1B, 2 and 3 | Day 1
  To assess the visual function
Pupillary function test in Part 2 | Up to week 8
  To assess the visual function
Pupillary function test in Part 1B and 3 | Day 1
  To assess the visual function
Full field stimulus threshold testing (FST) in Part 2 | Up to week 8
  To assess the visual function
FST in Part 1B | Day 1
  To assess the visual function

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Site JP00001, Meguro-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Fujinami-Yokokawa Y, Yang L, Joo K, Tsunoda K, Liu X, Kondo M, Ahn SJ, Li H, Park KH, Tachimori H, Miyata H, Woo SJ, Sui R, Fujinami K. Occult Macular Dysfunction Syndrome: Identification of Multiple Pathologies in a Clinical Spectrum of Macular Dysfunction with Normal Fundus in East Asian Patients: EAOMD Report No. 5. Genes (Basel). 2023 Sep 26;14(10):1869. doi: 10.3390/genes14101869. PMID 37895218